CLINICAL TRIAL: NCT01714193
Title: An Open-label Drug-Drug Interaction Study in Healthy Female Subjects to Explore the Effects of Multiple Doses of JNJ-28431754 on the Pharmacokinetics and Safety of Single Doses of an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel
Brief Title: A Study to Assess the Effects of Canagliflozin (JNJ-28431754) on the Pharmacokinetics and Safety of an Oral Contraceptive in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014755; 28431754DIA1002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Contraceptives, Oral; Ethinyl Estradiol; Levonorgestrel; LEVORA
MeSH Terms: interventions — Contraceptives, Oral; Ethinyl Estradiol-Norgestrel Combination; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin + oral contraceptive (Experimental): Each volunteer will receive a single dose of an oral contraceptive containing ethinyl estradiol and levonorgestrel on Day 1, followed by canagliflozin (JNJ-28431754) once daily on Days 4 through 8. On Day 9 volunteers will receive a single dose of an oral contraceptive containing ethinyl estradiol and levonorgestrel in combination with a single dose of canagliflozin.
  Interventions: Drug: Oral contraceptive; Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Oral contraceptive — One tablet (0.150 mg of levonorgestrel and 0.030 mg of ethinyl estradiol) taken orally (by mouth) on Day 1 and Day 9.
  Other Names: Levora
Drug: Canagliflozin (JNJ-28431754) — One 200 mg tablet taken orally (by mouth) on Days 4 through 9.
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to investigate whether there is a drug-drug interaction between multiple doses of canagliflozin (JNJ-28431754) and single doses of an oral contraceptive containing ethinyl estradiol and levonorgestrel. The safety and tolerability of canagliflozin will also be assessed in healthy volunteers.

DETAILED DESCRIPTION:
This study will be an open-label (all volunteers and study staff know the identity of the assigned treatment), single-center, fixed-sequence study (all volunteers receive the same medication on the same days), to determine how canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) affects the pharmacokinetics (ie, how the body affects the drug) of an oral contraceptive containing ethinyl estradiol and levonorgestrel. The study will consist of 3 phases; a screening phase, an open-label treatment phase, and an end-of-study (or follow-up) phase. Each volunteer will participate in the study for approximately 33 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer must have a body mass index (weight [kg]/height [m2]) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Volunteer must be a non-smoker (has not used tobacco or nicotine products in 6 months)

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* History of, or presence of, disorders commonly accepted as contraindications to sex hormonal therapy and contraindications to therapy with combined oral contraceptives
* Volunteer has used, or is currently using, any hormonal contraceptive within 30 days of admission to the study center or has received Depo Provera (or other combined contraceptive injection or hormonal contraceptive implant) in the 6 months prior to screening
* Volunteer is breast-feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of ethinyl estradiol and levonorgestrel | Up to Day 12
  Comparison of plasma concentrations of ethinyl estradiol and levonorgestrel, before and after administration of multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacokinetic interaction between multiple doses of canagliflozin and single doses of an oral contraceptive containing ethinyl estradiol and levonorgestrel.

SECONDARY OUTCOMES:
Plasma concentrations of canagliflozin (JNJ-28431754) | Days 8 and 9
  Comparison of plasma concentrations of canagliflozin (JNJ-28431754) before and after administration of a single dose of an oral contraceptive containing ethinyl estradiol and levonorgestrel. This will be used to determine whether there is a pharmacokinetic interaction between multiple doses of canagliflozin and single doses of an oral contraceptive containing ethinyl estradiol and levonorgestrel.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Vaccaro N, Bernard A, Skee D, Mamidi RN, Tian H, Weiner S, Stieltjes H, Sha S, Rothenberg P. Effect of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on the pharmacokinetics of oral contraceptives, warfarin, and digoxin in healthy participants. Int J Clin Pharmacol Ther. 2015 Jan;53(1):41-53. doi: 10.5414/CP202157. PMID 25345427